CLINICAL TRIAL: NCT02899104
Title: Current Management, Treatment Patterns and Outcomes of Metastatic Castrate Resistant Prostate Cancer Patients Treated With Radium-223
Brief Title: Navigant Study- Treatment Patterns in mCRPC (Metastatic Castrate Resistant Prostate Cancer )
Acronym: Navigant
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 18919
Record Dates: First submitted 2016-07-19; First posted 2016-09-14 (Estimated); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Prostatic Neoplasms, Castration-Resistant
MeSH Terms: conditions — Prostatic Neoplasms, Castration-Resistant | interventions — radium Ra 223 dichloride

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Radium-223 dichloride: Patients were diagnosed with bone metastatic castration-resistant prostate cancer (mCRPC), at least 18 years of age, must have received at least one intravenous injection of Radium-223.
  Interventions: Drug: Xofigo (Radium-223 dichloride, BAY88-8223)

INTERVENTIONS:
Drug: Xofigo (Radium-223 dichloride, BAY88-8223) — Xofigo is indicated for the treatment of patients with castration-resistant prostate cancer (CRPC), symptomatic bone metastases and no known visceral metastatic disease.

SUMMARY:
Categorize the clinical parameters and patient determinants that drive physician decision making for treatment selection including Radium-223 for patients with mCRPC.

DETAILED DESCRIPTION:
This is a chart review of 200 Xofigo patients to describe sequencing and characterize clinical parameters and patient determinants that drive physician decision making.

ELIGIBILITY:
Inclusion Criteria:

* Patients were diagnosed with bone metastatic castration-resistant prostate cancer (mCRPC) per medical chart.
* Patients were at least 18 years of age as of the first diagnosis for mCRPC.
* Patients must have received at least one intravenous injection of Radium-223 (Xofigo).
* First injection of Radium-223 must have started between periods

  1-January-2014 to 30-June-2014 or 15-November-2014 to present.
* Patients must have a minimum of 12 months documented follow-up records following last Radium-223 treatment or death within 12 months of last dose.

Exclusion Criteria:

* Patients who received Radium-223 as part in an interventional clinical trial
* Actively treated, or expect to be treated, in 6 months before last follow-up, for any other malignancy with the exception of non-metastatic skin cancer or low-grade superficial bladder cancer.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: mCRPC patients treated with Xofigo from 10 centers in the US
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Determining factors that drive physician decision for treatment selection. | Up to 9 months
  The treating physician should select out of the following options: Prostate Specific Antigen rising, Alkaline phosphatase (ALP) , Lactate dehydrogenase (LHD), testosterone, pain, symptoms, bone lesions, disease progression.

SECONDARY OUTCOMES:
Most common treatment sequences | Up to 9 months
  Description of what treatments are given to treat mCRPC in first, second, third, and fourth line.
Integration of Xofigo into the common treatment sequences, monotherapy or in combination. | Up to 9 months
  Describe where is Xofigo given in the treatment paradigm, whether is given in combination with hormonals or chemotherapy or given as a monotherapy
Mean Xofigo dose | Up to 9 months
  Mean dose of each treatment received in the respective sequence
Duration of Xofigo treatment | Up to 9 months
  Mean number of treatment cycles
Overall survival (OS) | Up to 9 months
  Collect outcomes for patients following treatment for mCRPC including changes in overall survival
Time to radiographic progression | Up to 9 months
  Collect outcomes for patients following treatment for mCRPC including changes in time to radiographic progression
Time to PSA (Prostate specific antigen) progression | Up to 9 months
  Collect outcomes for patients following treatment for mCRPC including changes in PSA progression
Most common SRE (Skeletal Related Event) | Up to 9 months
  The SRE occurring in the highest number of participants will be described.
Most common clinical intervention | Up to 9 months
  Most common clinical intervention to treat SRE/SSEs such as radiation or bone surgery.
Time to first SSE(Symptomatic Skeletal Events) | Up to 9 months
  Time to first SSE outcome will be analysed using the Kaplan Meier method
Reasons for discontinuation | Up to 9 months
  The treating physician should select out of the following options: Prostate Specific Antigen rising, Alkaline phosphatase (ALP) , Lactate dehydrogenase (LHD)), testosterone, pain, symptoms, bone lesions, disease progression.
Change in laboratory values from baseline | Up to 9 months
  for hemoglobin, platelets, neutrophils
Radiological progression free survival (rPFS) | Up to 9 months
  change in laboratory values from baseline for radiological progression free survival (rPFS)
Time to alkaline phosphatase (ALP) progression | Up to 9 months
  change in laboratory values from baseline for ALP
Time to visceral metastasis | Up to 9 months
  time from baseline to the appearance of visceral metastasis
Time to onset of first subsequent treatment | Up to 9 months
  or start of any other treatment for mCRPC
Pain | Up to 9 months
  Based on chart reported pain
Most common symptoms | Up to 9 months
  The participant and the treating physician should select out of the following list: fatigue, hypertension, cognitive disorder, seizures, edema, hypokalemia, cardiac disorders, hepatotoxicity, anemia, neutropenia, febrile neutropenia, thrombocytopenia
Type of physician | Up to 9 months
  Define type of physicians that treat of mCRPC
Change in PSA from baseline to 12 weeks, and baseline to discontinuation | Baseline and 12 weeks,Baseline and through study completion, an average of 1 year
  Measure PSA closed to the time of Xofigo initiation, 12 weeks after initiation and after discontinuation
Resource utilization | Up to 9 months
  Number of outpatient, inpatient and emergency room visits as well as number of hospitalizations
Change in ALP from baseline to 12 weeks, and baseline to discontinuation | Baseline and 12 weeks,Baseline and through study completion, an average of 1 year
  Measure ALP closed to the time of Xofigo initiation, 12 weeks after initiation and after discontinuation
Change in LDH from baseline to 12 weeks, and baseline to discontinuation | Baseline and 12 weeks,Baseline and through study completion, an average of 1 year
  Measure LDH values closed to the time of Xofigo initiation, 12 weeks after initiation and after discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Whippany, Whippany, New Jersey, United States

REFERENCES:
- See also: Related Info — http://clinicaltrials.bayer.com